CLINICAL TRIAL: NCT06668402
Title: Prospective Observational Study of the Association Between Daily Step Count and Treatment Response in Patients With Locally Advanced Rectal Cancer Undergoing Total Neoadjuvant Therapy: STEP-R Trial
Brief Title: Study of Daily Step Count and Treatment Response in Rectal Cancer (STEP-R)
Acronym: STEP-R
Status: Active, not recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Orhun Akdoğan, Principal Investigator, Gazi University
Other Study IDs: AESH-BADEK-2024-725
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Exercise; Total Neoadjuvant Treatment; Rectal Tumors; Smart Watch; Quality of Life (QOL)
MeSH Terms: conditions — Motor Activity; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Utilizing a smartwatch to gather data on individuals receiving treatment for rectal neoplasm. — Employing a smartwatch to monitor steps, sleep quality, intense physical activity, and vital signs in persons undergoing treatment for rectal carcinoma.

SUMMARY:
This study aims to examine the impact of daily physical activity, specifically step count, on treatment outcomes and side effects in patients with locally advanced rectal cancer receiving total neoadjuvant therapy (chemotherapy and radiotherapy before surgery). Using Huawei Watch Fit 2 smartwatches, we will track participants' daily step counts, heart rate, and sleep quality.

The primary hypothesis is that higher step counts and physical activity levels correlate with higher rates of complete pathological response at surgery. A secondary hypothesis is that increased physical activity may be associated with fewer or less severe side effects during treatment.

Participants will wear a smartwatch and complete the EORTC QLQ-C30 Quality of Life Questionnaire and the Pittsburgh Sleep Quality Index at the beginning and end of treatment. Data from the smartwatch, including step count, heart rate changes, and sleep duration, will be reviewed weekly during routine visits.

Approximately 200 patients with rectal cancer will participate, and each will be followed from the start of therapy until surgery (around 4-6 months). Total data collection is expected to take 12-15 months.

This study could improve cancer care by identifying links between physical activity and treatment outcomes, supporting future exercise guidelines for oncology patients.

DETAILED DESCRIPTION:
Background and Rationale Rectal cancer treatment includes a multimodal approach, often involving total neoadjuvant therapy (TNT), which combines chemotherapy and radiotherapy before surgical intervention. While physical activity, particularly walking, has shown general health benefits for cancer patients, the specific effects of objectively measured daily activity on treatment outcomes, such as response rates and side effect incidence, remain insufficient. Current methods for assessing physical activity largely rely on self-reported data, which can be less accurate. This study uses wearable technology (Huawei Watch Fit 2 smartwatches) to gather objective, real-time data on patients' physical activity, offering a novel approach to tracking exercise and health metrics throughout cancer treatment.

Study Objectives Primary Objective: To determine whether higher physical activity levels, specifically daily step counts, are associated with increased complete pathological response rates in rectal cancer patients undergoing TNT.

Secondary Objectives:

To evaluate the relationship between physical activity (step count) and the frequency and severity of treatment-related side effects.

To assess changes in sleep quality and heart rate as additional metrics of physical well-being and their potential influence on treatment tolerance and outcomes.

Methodology Participants: This study will include approximately 200 patients diagnosed with locally advanced rectal cancer and scheduled to begin TNT. Eligibility criteria focus on patients who can safely undergo physical activity monitoring and do not have contraindications for wearable device use.

Data Collection with Smartwatches:

Physical Activity: The smartwatch will track daily step counts and duration of physical activity that elevates the heart rate by at least 20% above the basal level.

Heart Rate Monitoring: Continuous heart rate data will be recorded to observe variability and detect any correlations with activity and side effect tolerance.

Sleep Quality: Sleep patterns and quality will be recorded to assess rest as a potential factor affecting treatment response.

Questionnaires: Two validated questionnaires will be administered:

EORTC QLQ-C30 (to assess cancer-related quality of life) and Pittsburgh Sleep Quality Index (to assess sleep quality and disturbances). Intervention and Monitoring Plan Weekly Monitoring: Patients will be seen weekly as part of their standard treatment schedule. During these visits, data from the smartwatch app (step count, heart rate, and sleep quality) will be reviewed alongside any updates on treatment side effects.

Duration and Follow-Up: Each participant will be followed from the initiation of TNT until surgical intervention (approximately 4-6 months). Data collection and follow-up are expected to span a total of 12-15 months for comprehensive data gathering across all enrolled patients.

Anticipated Outcomes and Significance This study aims to enhance understanding of physical activity's role in cancer treatment. By leveraging wearable technology to gather objective data, the study seeks to establish whether physical activity metrics correlate with treatment efficacy and side effect profiles. If successful, the findings could support integrating exercise recommendations into routine oncology care, tailored to individual patient metrics.

Future Directions Pending study outcomes, further research could focus on expanded trials in diverse cancer types, potentially using smartwatches to guide individualized exercise protocols, adjust treatment regimens, and support patient education on activity benefits during cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Diagnosed with locally advanced rectal cancer (stage II or III) and eligible for total neoadjuvant therapy (TNT).
* Planned to undergo chemotherapy and radiotherapy as part of neoadjuvant treatment before surgery.
* Capable of providing informed consent.
* Able to wear and operate the Huawei Watch Fit 2 smartwatch throughout the treatment period.
* Sufficient mobility to engage in physical activity, including walking, as per study requirements.
* Willing to complete weekly monitoring visits and complete the EORTC QLQ-C30 and Pittsburgh Sleep Quality Index questionnaires at baseline and study end

Exclusion Criteria:

* Stage I or metastatic (stage IV) rectal cancer.
* Contraindications to physical activity, including but not limited to severe cardiovascular or respiratory conditions that limit mobility.
* Prior treatment for rectal cancer with chemotherapy or radiotherapy.
* Use of a pacemaker or other implanted medical devices that might interfere with smartwatch functionality.
* Known allergic reaction to materials in the Huawei Watch Fit 2 smartwatch.
* Severe cognitive or psychological disorders that would hinder participation in the study or completion of questionnaires.
* Any medical or psychiatric condition that, in the opinion of the investigator, may compromise patient safety or interfere with study adherence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve adult patients diagnosed with locally advanced rectal cancer (stages II and III) who are scheduled to receive total neoadjuvant therapy (TNT), which includes chemotherapy and radiotherapy prior to surgery. Participants are required to have sufficient physical capacity for regular activity monitoring via a wearable smartwatch, which will collect data on physical activity, heart rate, and sleep quality. Stage I and metastatic (stage IV) rectal cancer patients are excluded, as they are not candidates for TNT. The study population represents individuals who are eligible for this preoperative treatment and can benefit from objective monitoring of activity as part of their treatment response assessment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The rate of pathological complete response in rectal cancer patients receiving neoadjuvant therapy | 9 months
  This outcome measure assesses the relationship between daily physical activity levels, specifically step count, and the rate of pathological complete response (pCR) in rectal cancer patients undergoing neoadjuvant therapy. By tracking patients' step counts throughout the treatment period, we aim to investigate whether higher physical activity levels correlate with a higher likelihood of achieving a pCR, defined as no residual tumor in resected tissue at the time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Yazici, Prof. Dr., Study Chair — Gazi University; Osman Sutcuoglu, Associate Professor, Study Director — Gazi University; Orhun Akdogan, MD, Principal Investigator — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital, Ankara, Yenimahalle
  - Gazi University, Ankara, Yenimahalle

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and in alignment with ethical guidelines protecting participant confidentiality. Data sharing is restricted to maintain compliance with institutional and national regulations governing patient privacy. Currently, no plans exist to provide IPD access beyond the research team responsible for the study.